CLINICAL TRIAL: NCT04986267
Title: The Effects of Hormonal Contraceptives on Incidence of ACL Injury Within Menstrual Cycle Phases
Status: Completed | Type: Observational
Sponsor: University of South Australia (Other)
Responsible Party: Principal Investigator, Tom Wycherley, Senior Lecturer in Exercise Science, University of South Australia
Other Study IDs: Buckley_2021
Record Dates: First submitted 2021-07-06; First posted 2021-08-02 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL Rupture: Female, aged 18-40 years of age with an acute ACL rupture of the knee that occurred within the last 3 months, who presented to a sports or orthopaedic clinic
  Interventions: Other: ACL Rupture

INTERVENTIONS:
Other: ACL Rupture — Female, aged 18-40 years of age with an acute ACL rupture of the knee that occurred within the last 3 months, who presented to a sports or orthopaedic clinic

SUMMARY:
The aim of this study is to investigate how hormonal contraceptives affect ACL rupture incidence within menstrual cycle phases. It is thought hormones such as estrogen and progesterone (which fluctuate throughout the normal menstrual cycle) play a role in the laxity of ligaments within the body. It is hypothesised that around the time of ovulation the ACL undergoes increased laxity, leaving it more likely to be injured. This study will look at the phase of the menstrual cycle in which the ACL injuries occur and whether there are differences due to the use and type of hormonal contraception participants may be using (such as Combined oral contraceptive, Mirena, Implanon), which can modify the levels of circulating estrogen and progesterone.

This study involves participants completing an anonymous electronic survey after presenting to a sports or orthopaedic clinic with an ACL rupture. The survey collects information about participant's current ACL injury and any previous knee injuries; typical menstrual cycle patterns and the use of hormonal contraception; and history of sports participation. Responses will be analysed to look for similarities and differences in ACL injury occurrence by menstrual cycle phase and hormonal contraceptive use.

The study hypotheses are:

1. Hormonal contraceptives that are known to reduce ovulatory rises in estrogen will have the most consistent pattern of ACL rupture incidence across all phases of the menstrual cycle.
2. There will be a mitigated risk of ACL rupture in the preovulatory phase of the menstrual cycle, relative to the other phases, in women using hormonal contraception compared to those not using hormonal contraception
3. There will be a higher proportion of ACL ruptures during the preovulatory phase of the menstrual cycle in non-hormonal contraceptive users.

DETAILED DESCRIPTION:
Anterior Cruciate ligament (ACL) rupture has been observed at higher rates in females than males during sporting competition, particularly during the preovulatory phase of the menstrual cycle. During the menstrual cycle, estrogen secretion varies from 10 to 100 fold throughout the cycle. A possible explanation for the ACL injuries being observed in the preovulatory phase, is that increases in estrogen levels increases the laxity of the ACL, predisposing it to risk of rupture. Studies investigating knee joint laxity, concluded that increased joint laxity was associated with an increased risk of ACL injury. In addition, measurement of knee laxity found no changes in laxity over time in males, but greater anterior displacement of the knee during the preovulatory phase of the menstrual cycle compared with the ovulatory and postovulatory phases in women.

Use of hormonal contraception typically maintains estradiol levels at ~25 pg/ml and decreases the ovulatory rise in estrogen. A study of the use of hormonal contraceptive in alpine skiers with ACL rupture reported that 74% of women were in the preovulatory phase (vs 26% in the postovulatory), experienced an ACL rupture. However, in women with ACL rupture in the preovulatory phase, 72.5% of the women were not using a hormonal contraceptive. A recent systematic review suggested an association between hormonal fluctuations and ACL injury and that hormonal contraceptives offer 20% reduction in risk of injury. Multiple modalities of hormonal and contraceptive control are available to females within Australia, but the efficacy of different hormonal contraceptives for reducing the risk of ACL rupture is unknown.

This study aims to investigate: 1) whether there are differences in risk of an ACL rupture incidence within menstrual cycle phases in females using different types of hormonal contraception. 2) whether there are differences in the pattern of ACL rupture incidence within menstrual cycle phases in females using vs not using hormonal contraception. 3) whether ACL rupture incidence in female athletes not using hormonal contraceptives are more prevalent during the pre-ovulatory phase of the menstrual cycle.

The study will use a cross-sectional design, with data being collected in women presenting at sports medicine or orthopaedic clinics with ACL rupture. On presentation at the clinic with ACL rupture, the study will be introduced to patients by a clinician and they will be shown a recruitment flyer that includes a QR code. On scanning the QR code patients will be taken to a RedCap survey website that they can enter an email in to receive, via automated reply email, a Participant Information Sheet and link to an anonymous study survey. The survey will take approximately 7 minutes to complete and asks questions about how the participants ACL injury occurred, any previous knee injuries, their menstrual cycle phase that the injury occurred in, their usual menstrual cycle characteristics, their use of hormonal contraceptives and the main sport they play.

Injury data will be analyzed according to menstrual cycle phase to confirm whether the preovulatory phase presents higher risk of ACL rupture than the ovulatory/postovulatory phase. Data will be stratified by hormonal contraception use and type to evaluate whether the injury occurrence pattern within the menstrual cycle differs by hormonal contraceptive use, such that the anticipated higher incidence in the preovulatory phase is mitigated with hormonal contraceptive use (and type).

The study hypotheses are:

1. Hormonal contraceptives that are known to reduce ovulatory rises in estrogen will have the most consistent pattern of ACL rupture incidence across all phases of the menstrual cycle.
2. There will be a mitigated risk of ACL rupture in the preovulatory phase of the menstrual cycle, relative to the other phases, in women using hormonal contraception compared to those not using hormonal contraception
3. There will be a higher proportion of ACL ruptures during the preovulatory phase of the menstrual cycle in non-hormonal contraceptive users.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to a sports or orthopaedic clinic with an acute ACL rupture of their knee that occurred within the last 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females who present to a sports or orthopaedic clinic with an ACL rupture that occurred within the previous 3 months
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
ACL Injury Menstrual Cycle Phase by Hormonal Contraceptive Type | Baseline
  In which phase of the menstrual cycle did the ACL injury occur, by hormonal contraceptive type (including non-use reference)

SECONDARY OUTCOMES:
ACL Injury Menstrual Cycle Phase by Hormonal Contraceptive Use | Baseline
  In which phase of the menstrual cycle did the ACL injury occur, by hormonal contraceptive use vs. non-use
ACL Injury Menstrual Cycle Phase Overall | Baseline
  In which phase of the menstrual cycle did the ACL injury occur (pooled group)

OTHER OUTCOMES:
ACL Injury Menstrual Cycle Phase, sensitivity analysis (Contact vs Non-Contact) | Baseline
  Examine robustness considering contact vs non contact injuries.
ACL Injury Menstrual Cycle Phase, sensitivity analysis (Previous knee injury) | Baseline
  Examine robustness considering previous serious knee injury (yes vs. no)
ACL Injury Menstrual Cycle Phase, sensitivity analysis (playing history/level) | Baseline
  Examine robustness considering player competition level
ACL Injury Menstrual Cycle Phase, sensitivity analysis (menstrual cycle status) | Baseline
  Examine robustness considering menstrual cycle status
ACL Injury Menstrual Cycle Phase, sensitivity analysis (menstrual cycle recall confidence) | Baseline
  Examine robustness considering menstrual cycle recall confidence
ACL Injury Menstrual Cycle Phase, sensitivity analysis (age) | Baseline
  Examine robustness considering age
ACL Injury Menstrual Cycle Phase, sensitivity analysis (BMI) | Baseline
  Examine robustness considering body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- UniSA Allied Health and Human Performance, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Data to be made available on request

REFERENCES:
- [Background] Fox A, Bonacci J, Hoffmann S, Nimphius S, Saunders N. Anterior cruciate ligament injuries in Australian football: should women and girls be playing? You're asking the wrong question. BMJ Open Sport Exerc Med. 2020 Apr 9;6(1):e000778. doi: 10.1136/bmjsem-2020-000778. eCollection 2020. PMID 32341803
- [Background] Renstrom P, Ljungqvist A, Arendt E, Beynnon B, Fukubayashi T, Garrett W, Georgoulis T, Hewett TE, Johnson R, Krosshaug T, Mandelbaum B, Micheli L, Myklebust G, Roos E, Roos H, Schamasch P, Shultz S, Werner S, Wojtys E, Engebretsen L. Non-contact ACL injuries in female athletes: an International Olympic Committee current concepts statement. Br J Sports Med. 2008 Jun;42(6):394-412. doi: 10.1136/bjsm.2008.048934. PMID 18539658
- [Background] Chidi-Ogbolu N, Baar K. Effect of Estrogen on Musculoskeletal Performance and Injury Risk. Front Physiol. 2019 Jan 15;9:1834. doi: 10.3389/fphys.2018.01834. eCollection 2018. PMID 30697162
- [Background] Ramesh R, Von Arx O, Azzopardi T, Schranz PJ. The risk of anterior cruciate ligament rupture with generalised joint laxity. J Bone Joint Surg Br. 2005 Jun;87(6):800-3. doi: 10.1302/0301-620X.87B6.15833. PMID 15911662
- [Background] Myer GD, Ford KR, Paterno MV, Nick TG, Hewett TE. The effects of generalized joint laxity on risk of anterior cruciate ligament injury in young female athletes. Am J Sports Med. 2008 Jun;36(6):1073-80. doi: 10.1177/0363546507313572. Epub 2008 Mar 7. PMID 18326833
- [Background] Deie M, Sakamaki Y, Sumen Y, Urabe Y, Ikuta Y. Anterior knee laxity in young women varies with their menstrual cycle. Int Orthop. 2002;26(3):154-6. doi: 10.1007/s00264-001-0326-0. Epub 2002 Apr 5. PMID 12073107
- [Background] Mishell DR Jr, Thorneycroft IH, Nakamura RM, Nagata Y, Stone SC. Serum estradiol in women ingesting combination oral contraceptive steroids. Am J Obstet Gynecol. 1972 Dec 1;114(7):923-8. doi: 10.1016/0002-9378(72)90098-1. PMID 4645131
- [Background] Wojtys EM, Huston LJ, Boynton MD, Spindler KP, Lindenfeld TN. The effect of the menstrual cycle on anterior cruciate ligament injuries in women as determined by hormone levels. Am J Sports Med. 2002 Mar-Apr;30(2):182-8. doi: 10.1177/03635465020300020601. PMID 11912085
- [Background] Beynnon BD, Shultz SJ. Anatomic alignment, menstrual cycle phase, and the risk of anterior cruciate ligament injury. J Athl Train. 2008 Sep-Oct;43(5):541-2. doi: 10.4085/1062-6050-43.5.541. No abstract available. PMID 18833305
- [Background] Herzberg SD, Motu'apuaka ML, Lambert W, Fu R, Brady J, Guise JM. The Effect of Menstrual Cycle and Contraceptives on ACL Injuries and Laxity: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2017 Jul 21;5(7):2325967117718781. doi: 10.1177/2325967117718781. eCollection 2017 Jul. PMID 28795075